CLINICAL TRIAL: NCT01975155
Title: Dietary Assessment and Mycotoxin Exposure in Celiac Subjects
Brief Title: Dietary Assessment and Mycotoxin Exposure in Celiac Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Parma (Other)
Responsible Party: Principal Investigator, Leda Roncoroni, Biologist, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 852/12; GFD/2012 (Other: Fondazione IRCCS Cà Granda administration)
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Gluten free diet nutrient content; mycotoxins; Gluten free diet
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine

GROUPS / COHORTS (2):
- Celiac: patients with celiac disease filling the questionnaire and undergoing urinary test
  Interventions: Other: food questionnaire; Other: Urinary mycotoxin test
- healthy controls: healthy patients filling the questionnaire and undergoing urinary test
  Interventions: Other: food questionnaire; Other: Urinary mycotoxin test

INTERVENTIONS:
Other: food questionnaire
Other: Urinary mycotoxin test

SUMMARY:
Celiac disease (CD) is the most common autoimmune enteropathy in Western Countries. Gluten free diet is the only available therapy but few is known about its nutrient content and mycotoxin exposure.

DETAILED DESCRIPTION:
Celiac disease (CD) is the most common autoimmune enteropathy in Western Countries, occurring in genetically susceptible individuals, elicited by the gluten ingestion. By definition the disease responds to gluten withdrawal, so currently gluten free (GFD) diet is the therapy for celiac patients. It is known that gluten rich products are important source of nutrients on the other hands it is not clear if gluten exclusion from the diet could have a negative effect on the nutritional status of CD patients.

Another concern related to the GFD could be the high exposure to mycotoxins due to the high concentration of maize in GF products.

AIM The aim of this study is to estimate the nutrient intake and the dietary exposure of all mycotoxin types in a group of treated celiac patients vs. non-celiac subjects.

METHODS We will enroll celiac patients and healthy controls. Exclusion criteria for celiac patients will be: 1) diagnosis of CD less than two years 2) age under 18 or over 70 3) associated metabolic or chronic disease 4) pregnancy or lactation 5) being vegetarian or vegan. Exclusion criteria for the healthy subjects will be the same with the exception of the diagnosis of CD.

Total food and beverage consumption will be assessed by means of a 7 days long questionnaire. All participants will be trained by a nutritionist to record all food consumed and the completed forms will be returned and reviewed during a face-to-face interview at which portions size were quantified in standard units. Participants will be asked to weigh all foods and drinks consumed and to provide a detailed description of each food, including methods of preparation and recipes, whenever possible. In case of Gluten Free Foods, patients will be asked to precisely note the name of the manufacturer or to provide the food label.

The nutrient intake was calculated using a software application linked to the food database of the European Institute of Oncology integrated with the nutrient composition of 60 commercial GF foods. The computer output will consist in the evaluation of the mean daily intake of macro nutrients for each subject, in terms of carbohydrates, protein and lipid. Food items consumed will be also collapsed into food categories; pasta, bread, potatoes, flours, different cereals, fruit, vegetables, milk, cheese, eggs, fish, oils and fats, biscuits, sweet snacks, breakfast cereals, candies, chocolate, soft drinks, juices, coffees, teas, alcoholic beverages. For each subject, the mean daily intake of each food category will be calculated.

The 24-h urines were collected at the end of the registration period and analyzed for mycotoxins.

ELIGIBILITY:
Inclusion Criteria:

* celiac disease diagnosis
* GFD for at least 2 years

Exclusion Criteria:

* follow a vegetarian diet
* being affected by important systemic or psychiatric disorders
* incapacity to fill the questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult subjects with or without celiac disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Mycotoxins | mycotoxins will be measured at the end of a 7 day period and the completion of the dietary questionnaire
  Urinary measure of mycotoxins

SECONDARY OUTCOMES:
dietary questionnaire | 7 days
  during a 7 days lonf period the patients will be invited to fill a complete dietary questionnaire on the basis of the questionnaire results the nutritional status will be evaluated At the end of these 7 days the patients will collect the 24h urine for mycotoxin dosage

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, MD, Study Chair — Celiac Disease Center, Fondazione IRCCS Cà Granda; Nicoletta Pellegrini, Study Chair — University of Parma; Dario Conte, MD, Study Chair — Celiac Disease Center, Fondazione IRCCS Cà Granda
Locations (1):
- Celiac Disease Center, Fondazione IRCCS Cà Granda, Milan, Italy

REFERENCES:
- [Derived] Morreale F, Agnoli C, Roncoroni L, Sieri S, Lombardo V, Mazzeo T, Elli L, Bardella MT, Agostoni C, Doneda L, Scricciolo A, Brighenti F, Pellegrini N. Are the dietary habits of treated individuals with celiac disease adherent to a Mediterranean diet? Nutr Metab Cardiovasc Dis. 2018 Nov;28(11):1148-1154. doi: 10.1016/j.numecd.2018.06.021. Epub 2018 Jul 4. PMID 30143412
- [Derived] Mazzeo T, Roncoroni L, Lombardo V, Tomba C, Elli L, Sieri S, Grioni S, Bardella MT, Agostoni C, Doneda L, Brighenti F, Pellegrini N. Evaluation of a Modified Italian European Prospective Investigation into Cancer and Nutrition Food Frequency Questionnaire for Individuals with Celiac Disease. J Acad Nutr Diet. 2016 Nov;116(11):1810-1816. doi: 10.1016/j.jand.2016.04.013. Epub 2016 May 28. PMID 27245762